CLINICAL TRIAL: NCT00962078
Title: Effects of a Complex Pulmonary Rehabilitation Program on Patients With End Stage Lung Diseases Undergoing Evaluation for Lung Transplantation (Pre-LTx)
Brief Title: Pulmonary Rehabilitation in Patients Before Lung Transplantation (LTx)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Dr, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRÄ-LTX-08022; Ethikkommission; Landesärztekammer Bayern; Nr. 08022
Record Dates: First submitted 2009-07-27; First posted 2009-08-19 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: COPD; Pre-Lung-Transplantation; Hypercapnia; Respiratory Insufficiency
Keywords: COPD; Pre-Lung-Transplantation; Intervall versus continuous training; 6 MWD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia; Respiratory Insufficiency | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interval training (Other): interval training in lung transplant candidates
  Interventions: Other: interval training
- Continuous Training (Other): continuous training in lung transplant candidates
  Interventions: Other: continuous endurance training

INTERVENTIONS:
Other: continuous endurance training — at 60 percent of peak Watt
  Arms: Continuous Training
Other: interval training — at 100 percent of peak Watt
  Arms: interval training

SUMMARY:
The purpose of this study is to study the effects of a complex pulmonary rehabilitation program on mobility measured by 6 minute walking distance (6MWD) and physical activity, measured via Dynaport and Actibelt Aktivitätsmonitor, dyspnoea (VAS), quality of life (HRQL (SF36, EuroQul)), anxiety and depression (HADS)and PaCO2-behavior under physical activity.

ELIGIBILITY:
Inclusion Criteria:

* pre-LTx (listed for lung-transplantation or currently undergoing evaluation)
* COPD Stadium IV GOLD
* α-1-Antitrypsin-deficiency-Emphysema
* respiratory Insufficiency
* oxygen therapy (LTOT)

Exclusion Criteria:

* serious Exacerbation (Symptoms longer than three days, change of therapy, e.i. antibiotics, steroids) during the last four weeks before rehabilitation
* clinical signs of manifest heart insufficiency
* acute coronar syndrome
* left heart insufficiency(EF < 40%)
* missing Compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Dr.med., Study Director — Klinikum Berchtesgadener Land, Schön-Kliniken
Locations (1):
- Klinikum Berchtesgadener Land, Schönau am Königssee, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interval Training | Continuous Training
Started | 35 | 36
Completed | 30 | 30
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interval Training | Continuous Training | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (6) | 55 (7) | 54 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  Germany | 36 | 35 | 71
FEV1% [Mean (Standard Deviation); unit: % predicted] | 24 (8) | 27 (7) | 25 (8)

OUTCOME MEASURES:

1. Primary Outcome: Effects of a Multimodal Pulmonary Rehabilitation Program on 6 Minute Walking Distance (6MWD)
Time Frame: value at day 21 minus value at day 1
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Interval Training | Continuous Training
Number analyzed (Participants) | 30 | 30
meter | 35 (29) | 36 (42)

2. Secondary Outcome: Dyspnoea During Exercise Measured on the Borg Scale
Description: The Borg scale is a numeric scale that ranges from 0 to 10 points to rate dyspnea.
  The scale is like follows:
  0 Nothing at all
  1. Very slight
  2. Slight
  3. Moderate
  4. Somewhat severe
  5. Severe
  7 Very severe 8 9 Very, very severe (almost maximal) 10 Maximal
Time Frame: mean values from day 1 to day 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interval Training | Continuous Training
Number analyzed (Participants) | 30 | 30
units on a scale | 6.2 (1.6) | 7.2 (1.4)

ADVERSE EVENTS:
Arm/Group | Interval Training | Continuous Training
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes